CLINICAL TRIAL: NCT02059577
Title: Nutritional and Dietary Treatment Study for Children/Adults With Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Autism Research Instittute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NutritionDietAutism
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Autism
Keywords: vitamins; minerals; essential fatty acids; Epsom salts; carnitine; digestive enzymes; gluten-free casein-free diet
MeSH Terms: conditions — Autistic Disorder | interventions — Diet Therapy; Vitamins; Fatty Acids, Essential; Carnitine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): This group received a combination of nutritional treatments, added sequentially, including vitamins/minerals, essential fatty acids, Epsom salt baths, carnitine, digestive enzymes, and healthy, gluten-free, casein-free diets.
  Interventions: Dietary Supplement: Nutritional and Dietary Interventions
- Non-Treatment Group (No Intervention): This group did not have any significant changes in their treatments for 12 months

INTERVENTIONS:
Dietary Supplement: Nutritional and Dietary Interventions — Day 0: Vitamin/Mineral supplementation begins. Day 30: Essential Fatty Acid supplementation begins. Day 60: Epsom Salt baths begin (2x/week) Day 90: Carnitine supplementation begins Day 180 Digestive Enzyme supplementation begins; Day 210: Healthy, casein-free, gluten-free diet is begun.
  Other Names: vitamin/mineral supplement; essential fatty acids; Epsom salt bath; carnitine; digestive enzymes; healthy gluten-free casein-free diet
  Arms: Treatment Group

SUMMARY:
70 children and adults with autism spectrum disorders will be enrolled in a 1-year, single-blind treatment study. Assessments will be conducted at the beginning and end of the study, including measurements of nutritional, metabolic, and digestive status and assessments of autism severity and overall functioning. Half of the participants will be randomized into a treatment study, and half will be randomized to no changes in their current treatments. Treatments will be added in a sequential manner over 12 months, including vitamin/minerals, essential fatty acids, carnitine, digestive enzymes, and healthy, gluten-free, casein-free diets. A dedicated team of nutritionists, nurses, and physicians will support and monitor the participants throughout the study.

A group of 50 neurotypical children and adults, of similar age and gender, will be included for comparison.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria - Autism Group

1. Diagnosis of autism spectrum disorder (autism, PDD-NOS, or Asperger's) by a psychiatrist, psychologist, or developmental pediatrician
2. Verification of diagnosis by an ADOS evaluation (conducted by ASU staff)
3. Age of 2.5 years to 60 years

Enrollment Criteria - Non-autism Group

1. No diagnosed mental disorders, including autism spectrum disorders, ADHD, depression, anxiety, etc.
2. No first-degree relatives of individuals with autism (no siblings or parents)
3. Age of 2.5 years to 60 years -

Exclusion Criteria:

Exclusion Criteria - Autism Group

1. Major changes in behavioral or medical treatments in the previous two months, or intention to make such changes during the 12 months of the study.
2. Usage of nutritional supplements (vitamins, minerals essential fatty acids, carnitine) or special diets in the previous two months

Exclusion Criteria - Non-autism Group 1) Usage of nutritional supplements (vitamins, minerals essential fatty acids, carnitine) or special diets in the previous two months

-

Ages: 30 Months to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2011-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Childhood Autism Rating Scale | 12 months
  Pre and post assessment of autism symptoms/severity
Reynolds Intellectual Assessment Scales | 12 months
  Pre and post test of intellectual ability
Vineland Adaptive Behavior Scale | 12 months
  Pre and post evaluation of adaptive behaviors

CONTACTS AND LOCATIONS:
Overall Officials: James B. Adams, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Tempe, Arizona, United States